CLINICAL TRIAL: NCT03943667
Title: A Phase III Randomized Study Evaluating Gemcitabine and Paclitaxel Versus Gemcitabine Alone After FOLFIRINOX Failure or Intolerance in Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Gemcitabine and Paclitaxel vs Gemcitabine Alone After FOLFIRINOX Failure in Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: GEMPAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0110/1809; 2018-002886-21 (EudraCT Number); PRODIGE 65 - UCGI 36 (Other: UNICANCER)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Metastatic Pancreas Ductal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GEMPAX (Experimental): Gemcitabine + Paclitaxel until progression
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel
- Control (Active Comparator): Gemcitabine alone until progression
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m² in IV infusion over 30-40 minutes at Day 1, 8 and 15 followed by one week of rest.
  Other Names: GEMZAR
Drug: Paclitaxel — 80 mg/m² in IV infusion over 60 minutes at Day 1, 8 and 15 followed by 1 week of rest.
  Other Names: TAXOL
  Arms: GEMPAX

SUMMARY:
This study aims to evaluate whether the combination of gemcitabine and paclitaxel allows to improve the overall survival compared to gemcitabine alone, in patients with metastatic Pancreatic Ductal Adenocarcinoma (PDAC) after FOLFIRINOX failure or intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Pancreatic Ductal Adenocarcinoma with histological or cytological proof
* Age ≥18 years
* At least 1 evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 outside any previously irradiated area
* Failure of first line FOLFIRINOX (Progressive disease during therapy of within 3 months +/- 15 days)
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
* Life expectancy ≥12 weeks
* Negative serology (HIV, hepatitis B and C)
* Adequate organs function
* Proven Post-menopausal status or negative urinary or serum pregnancy test
* Woman of childbearing potential and male patients must agree to use adequate contraception fo the duration of the trial and up to 6 months after completing treatment
* Patients affiliated to the social security system
* Patient must have signed a written informed consent form

Exclusion Criteria:

* Any other primary tumor or secondary malignancy except basal cell carcinoma of skin or in situ carcinoma of the cervix uteri
* Known cerebral metastasis
* Uncontrolled severe infections
* Patients with Kaposi's sarcoma
* Peripheral neuropathy exceeding grade 2 on Common Terminology Criteria for Adverse Events (CTCAE) v5.0
* Previous treatment with taxane and/or gemcitabine (for pancreas cancer only)
* Patients with known allergy or severe hypersensitivity to any trial drug or drug excipient
* Patients with any other disease or illness which requires hospitalisation or is incompatible with the trial treatment
* Patients unable to comply with trial obligations for geographic, social or physical reasons, or who are unable to understand the purpose and procedures of the trial
* Participation in another clinical trial within 14 days prior to randomization
* Patients deprived of liberty or under legal protection measures or patients whose willingness to participate in the trial may be unduly influenced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle de la FOUCHARDIERE, Dr, Principal Investigator — UNICANCER
Locations (26):
- France (26):
  - CH de Bayeux, Bayeux
  - CH Simone Veil, Beauvais
  - CHU Jean Minjoz, Besançon
  - Hôpital Duchenne, Boulogne-sur-Mer
  - CH du Cotentin, Cherbourg
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hospices civils de Lyon, Lyon
  - CHU La Timone, Marseille
  - Hôpital Européen de Marseille, Marseille
  - Hôpital Saint-Joseph, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Nord Franche Comté, Montbéliard
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint-Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Rouen, Rouen
  - Institut Curie, Saint-Cloud
  - CHU de Saint-Etienne, Saint-Etienne
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Hôpital Broussais, St-Malo
  - Hôpital Trousseau, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Derived] De La Fouchardiere C, Malka D, Cropet C, Chabaud S, Raimbourg J, Botsen D, Launay S, Evesque L, Vienot A, Perrier H, Jary M, Rinaldi Y, Coutzac C, Bachet JB, Neuzillet C, Williet N, Desgrippes R, Grainville T, Aparicio T, Peytier A, Lecomte T, Roth GS, Thirot-Bidault A, Lachaux N, Bouche O, Ghiringhelli F. Gemcitabine and Paclitaxel Versus Gemcitabine Alone After 5-Fluorouracil, Oxaliplatin, and Irinotecan in Metastatic Pancreatic Adenocarcinoma: A Randomized Phase III PRODIGE 65-UCGI 36-GEMPAX UNICANCER Study. J Clin Oncol. 2024 Mar 20;42(9):1055-1066. doi: 10.1200/JCO.23.00795. Epub 2024 Jan 17. PMID 38232341

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GEMPAX | Control
Started | 140 | 71
Completed | 140 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GEMPAX | Control | Total
Number analyzed (Participants) | 140 | 71 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 36 | 106
  >=65 years | 70 | 35 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 28 | 81
  Male | 87 | 43 | 130
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 140 | 71 | 211

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from the date of randomization to the date of death from any cause
Time Frame: Until death (life expectancy around 12 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GEMPAX | Control
Number analyzed (Participants) | 140 | 71
months | 6.4 [5.2 to 7.4] | 5.9 [4.6 to 6.9]

ADVERSE EVENTS:
Time Frame: GEMPAX tracks adverse events for each participant from their first treatment dose, at day 1, day 8 and day 15 of each treatment cycle, and up to 30 days after the day of last treatment dose, approximatively 7 months.
Arm/Group | GEMPAX | Control
All-Cause Mortality (participants affected / at risk) | 131/140 | 68/71
Serious Adverse Events (participants affected / at risk) | 71/140 | 26/71
Other Adverse Events (participants affected / at risk) | 138/140 | 22/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEMPAX (N=140) | Control (N=71)
ANAEMIA (Blood and lymphatic system disorders) | 7 | 1
BICYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0
CARDIAC FAILURE (Cardiac disorders) | 2 | 0
APLASIA (Congenital, familial and genetic disorders) | 1 | 1
VISION BLURRED (Eye disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 2
ANASTOMOTIC ULCER PERFORATION (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7 | 2
MELAENA (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
SUBILEUS (General disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 4 | 0
ASTHENIA (General disorders) | 1 | 0
GENERA PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 2
HYPERTHERMIA (General disorders) | 1 | 0
HYPOTHERMIA (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
PYREXIA (General disorders) | 3 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 | 1
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 2 | 3
CHOLANGITIS (Hepatobiliary disorders) | 4 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITITS ACUTE (Hepatobiliary disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 2
BACTERAEMIA (Infections and infestations) | 1 | 0
BILIARY SEPSIS (Infections and infestations) | 1 | 0
BILIARY TRACT INFECTION (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1
INJECTION SITE INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 1
SEPSIS (Infections and infestations) | 1 | 1
VASCULAR ACCESS SITE INFECTION (Infections and infestations) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
STARVATION (Metabolism and nutrition disorders) | 1 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
COMA (Nervous system disorders) | 1 | 0
DYSKINESIA (Nervous system disorders) | 1 | 0
HYPERAESTHESIA (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
PSYCHOMOTOR SKILLS IMPAIRED (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEMPAX (N=140) | Control (N=71)
ANAEMIA (Blood and lymphatic system disorders) | 21 | 3
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 22 | 11
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 20 | 3
CARDIAC FAILURE (Cardiac disorders) | 2 | 0
APLASIA (Congenital, familial and genetic disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
STOMATITIS (Gastrointestinal disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
ASTHENIA (General disorders) | 14 | 2
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 3 | 0
CHOLESTASIS (Hepatobiliary disorders) | 1 | 0
HEPATIC CYTOLISIS (Hepatobiliary disorders) | 4 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 0
PLATELET COUNT DECREASED (Investigations) | 7 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 17 | 0
NEUROTOXICITY (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0
PERIPHERAL SENSORY NEUTROPATHY (Nervous system disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
INTERSITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 | 0
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03943667/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03943667/SAP_001.pdf